CLINICAL TRIAL: NCT01453569
Title: Phase II Study of Sodium Oligo-mannurarate Capsule on Mild to Moderate Alzheimer Disease
Brief Title: Safety, Efficacy and Dose Titration of Sodium Oligo-mannurarate Capsule on Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Greenvalley Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9712011-1
Record Dates: First submitted 2011-09-30; First posted 2011-10-18 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- sodium oligo-mannurarate 900mg (Experimental)
  Interventions: Drug: Sodium oligo-mannurarate 900mg
- sodium oligo-mannurarate 600mg (Experimental)
  Interventions: Drug: Sodium oligo-mannurarate 600mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium oligo-mannurarate 600mg — sodium oligo-mannurarate capsule 600mg twice a day for 24 weeks
  Other Names: Sodium oligo-mannurarate low dose
  Arms: sodium oligo-mannurarate 600mg
Drug: Sodium oligo-mannurarate 900mg — sodium oligo-mannurarate capsule 900mg twice a day for 24 weeks
  Other Names: Sodium oligo-mannurarate high dose
  Arms: sodium oligo-mannurarate 900mg
Drug: Placebo — simulant of sodium oligo-mannurarate capsule
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether sodium oligo-mannurarate capsule is effective and safe in the treatment of mild to moderate alzheimer' disease, and to determine the best therapeutic dose of sodium oligo-mannurarate capsule.

DETAILED DESCRIPTION:
Alzheimer's disease is known for placing a great burden on caregivers which includes social, psychological, physical or economic aspects. Research indicates that the disease is associated with plaques and tangles in the brain. Currently used treatments offer a small symptomatic benefit. No treatments to delay or halt the progression of the disease are, as of yet, available. The investigators suppose sodium oligo-mannurarate capsule to be effective to halt the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* At least primarily educated.
* Accord with Probable Alzheimer disease of National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association(NINCDS-ADRDA)'s Criteria.
* 10 points ≤ Minimum Mean-Square Error(MMSE) ≤ 24 points.
* Hachinski ischemia scale <4 points.
* Hamilton depression scale ≤10 points.
* Should have stable accompanying person, or at least contact 2 hours per day, 4 days per week with accompanying person. The accompanying person should help the patient throughout the trial.
* Signed the information consent form.

Exclusion Criteria:

* Have been in other clinical trials within 30 days before this trial' start.
* women during pregnancy or lactation.
* Dementia caused by other diseases.
* previous nervous system diseases.
* Abnormal laboratory results.
* Uncontrolled hypertension.
* Unstable or serious diseases of heart, lung, liver, kidney and blood.
* Visual or auditory handicap.
* Significant focal lesions revealed by electronic computer X-ray tomography(CT) or magnetic resonance imaging(MRI) in one year before enrollment.
* Alcohol abuse or drug abuse.
* psychotic, including patients with serious depression.
* Patients being in drug therapy of Alzheimer disease which cannot be stopped.
* In treatment of heparin, Polysaccharide sulfate, mannose ester 3 weeks before the recruitment.
* Investigator consider the patient cannot finish this trial for any reason.
* Relatives or employees of the investigators, staff of the investigate centers, contract research organization and sponsor.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shifu Xiao, M.D., Principal Investigator — Shanghai Mental Health Center
Locations (24):
- China (24):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing Medical University Second Affiliated Hospital, Chongqing, Chongqing Municipality
  - The First Affliated Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - The Third Affliated Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Brain Hospital, Guangzho, Guangdong
  - The 251 Hospital of People's Liberation Army, Zhangjiakou, Hebei
  - The First Affliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Wuhan General Hospital of Guangzhou Military of People's Military Army, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Central Hospital of Baotou, Baotou, Inner Mongolia
  - The Affliated Brain Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - The First Affliated Hospital of Chinese Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - The Ninth Hospital, Shanghai Jiao Tong University school of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center , Shanghai Jiao Tong University school of Medicine, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Forth Military Medical University of PLA, Xi’an, Shanxi
  - West China Hospital, West China School of Medicine Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Medical college of Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wang T, Kuang W, Chen W, Xu W, Zhang L, Li Y, Li H, Peng Y, Chen Y, Wang B, Xiao J, Li H, Yan C, Du Y, Tang M, He Z, Chen H, Li W, Lin H, Shi S, Bi J, Zhou H, Cheng Y, Gao X, Guan Y, Huang Q, Chen K, Xin X, Ding J, Geng M, Xiao S. A phase II randomized trial of sodium oligomannate in Alzheimer's dementia. Alzheimers Res Ther. 2020 Sep 14;12(1):110. doi: 10.1186/s13195-020-00678-3. PMID 32928279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo
Started | 86 | 84 | 85
Completed | 75 | 70 | 78
Not Completed | 11 | 14 | 7

BASELINE CHARACTERISTICS:
Population: All the treated subjects were evaluated for safety. 2, 8 and 3 subjects were excluded from FAS in placebo, 600 mg and 900 mg group respectively. So the case No. were 83, 76, 83 for placebo, 600 mg and 900 mg group respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo | Total
Number analyzed (Participants) | 83 | 76 | 83 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.39 (8.51) | 70.26 (8.40) | 70.34 (8.13) | 70.33 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 41 | 52 | 143
  Male | 33 | 35 | 31 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change of Alzheimer's Disease Assessment Scale-cognitive Subscale(ADAS-cog)/12 After 24 Wks Treatment of Sodium Oligo-mannurarate Capsule
Description: Alzheimer's Disease Assessment Scale-cognitive Subscale(ADAS-cog)/12 is the most popular cognitive testing instrument used in clinical trials. It consists of 12 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities which are often referred to as the core symptoms of AD. The total score ranges 0-75, the higher score indicates more severity of the disease. Change after 24 wks treatment was calculated by the week 24 minus week 0 (baseline), and a negative change represents an improvement.
Time Frame: 24 weeks
Population: 85, 84, 86 patients were enrolled, and 2, 8 and 3 subjects were excluded from FAS in placebo, 600 mg and 900 mg group respectively. So the case No. ananlysed were 83, 76, 83 for placebo, 600 mg and 900 mg group respectively.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo
Number analyzed (Participants) | 83 | 76 | 83
units on a scale | -2.58 (0.62) | -1.39 (0.75) | -1.45 (0.77)

2. Secondary Outcome: Change of Clinician's Interview-Based Impression of Change Plus(CIBIC-plus) After 24 Wks Treatment of Sodium Oligo-mannurarate Capsule
Description: Clinician's Interview-Based Impression of Change Plus(CIBIC-plus) is widely used in antidementia drug trials. It comprises Likert scales for disease severity and changes, and written accounts summarizing semistructured interviews evaluating behavior, cognition, and function. The results classified as 7 degrades as: Markedly improved, Moderately improved, Minimally improved, No change, Minimally worse, Moderately worse, and Markedly worse.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo
Number analyzed (Participants) | 83 | 76 | 83
participants
  Markedly improved | 0 | 2 | 3
  Moderately improved | 13 | 9 | 6
  Minimally improved | 29 | 18 | 32
  No change | 35 | 23 | 25
  Minimally worse | 4 | 21 | 17
  Moderately worse | 2 | 3 | 0
  Markedly worse | 0 | 0 | 0

3. Secondary Outcome: Change of Alzheimer's Disease Cooperative Study/Activities of Daily(ADCS-ADL) After 24 Wks Treatment of Sodium Oligo-mannurarate Capsule
Description: Alzheimer's Disease Cooperative Study/Activities of Daily (ADCS-ADL) is a scale assessed the daily activties of AD patients after interviewed the caregiver. The scale mainly assess the eating, walking, writing, bathing and reading, et al of the subject. The total score ranges 0-78, the higher score indicate improvement in daily activities. Change after 24 wks treatment was calculated by the week 24 minus week 0 (baseline), and a positive change represents an improvement.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo
Number analyzed (Participants) | 83 | 76 | 83
units on a scale | -0.49 (0.91) | -0.47 (0.88) | -1.06 (0.85)

4. Secondary Outcome: Change of Neuropsychiatric Inventory(NPI) After 24 Wks Treatment of Sodium Oligo-mannurarate Capsule
Description: Neuropsychiatric Inventory (NPI) is a scale to obtain information on the presence of psychopathology in patient with brain disorders. The NPI was developed for application to patients with AD and other dementias, but it may be useful in the assessment of behavioral changes in other conditions. Twelve behavioral areas included in the NPI will be assessed in this trial: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety and elation/euphoria, et al. The total score ranges 0 to 120, the higher score indicates worse state of the AD patient. Change after 24wks treatmnt was calculated by the week 24 minus week 0 (baseline), and a negative change represents an improvement.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo
Number analyzed (Participants) | 83 | 76 | 83
units on a scale | -1.11 (1.22) | 0.24 (0.83) | -2.08 (0.98)

ADVERSE EVENTS:
Arm/Group | Sodium Oligo-mannurarate 900mg | Sodium Oligo-mannurarate 600mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/86 | 6/84 | 6/85
Other Adverse Events (participants affected / at risk) | 3/86 | 12/84 | 5/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oligo-mannurarate 900mg (N=86) | Sodium Oligo-mannurarate 600mg (N=84) | Placebo (N=85)
Behavioral and psychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Subdural hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Implantation of artificial heart pacemaker (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paralysis of oculomotor nerve (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Emptying disorder of intestine and stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chill (General disorders) | 0 (0) | 0 (0) | 1 (1)
Compressive fracture of vertebra (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oligo-mannurarate 900mg (N=86) | Sodium Oligo-mannurarate 600mg (N=84) | Placebo (N=85)
Ear and labyrinth (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) — Medication-related AE
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) — Medication-related AE
Injuries, toxicosis, complications due to surgery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Medication-related AE
Muscular and connective tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Medication-related AE
CNS disorders (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Medication-related AE
Psychiatiric disorders (Psychiatric disorders) | 0 (0) | 5 (5) | 0 (0) — Medication-related AE
Reproductive system and mammary gland (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Medication-related AE
Respiratoty system, chest and mediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Medication-related AE
Dermatologic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) — Medication-related AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other